CLINICAL TRIAL: NCT00939848
Title: Randomised Phase II Trial of Cediranib (AZD2171) Versus Placebo in Addition to Cisplatin/Gemcitabine Chemotherapy for Patients With Advanced Biliary Tract Cancers
Brief Title: Cediranib Versus Placebo Plus Cisplatin/Gemcitabine Chemotherapy for Patients With Advanced Biliary Tract Cancers
Acronym: ABC-03
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABC-03 09/0193
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2012-10

CONDITIONS: Biliary Tract Neoplasms
Keywords: Disease-Free Survival
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; cediranib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): The experimental arm will consist of cisplatin 25 mg/m2 plus gemcitabine 1000 mg/m2 on days 1 and 8 of a 21-day cycle with cediranib 20mg oral daily (continuous dosing).
  Interventions: Drug: cisplatin; Drug: cediranib; Drug: gemcitabine
- Arm A (Placebo Comparator): The control arm will consist of cisplatin 25 mg/m2 plus gemcitabine 1000 mg/m2 on days 1 and 8 of a 21-day cycle with a matching placebo 20mg oral daily (continuous dosing)
  Interventions: Drug: gemcitabine; Drug: cisplatin; Drug: Placebo

INTERVENTIONS:
Drug: gemcitabine — gemcitabine 1000 mg/m2 on days 1 and 8 of a 21-day cycle for 24 weeks in the absence of disease progression
  Arms: Arm A
Drug: cisplatin — cisplatin 25 mg/m2 on days 1 and 8 of a 21-day cycle for 24 weeks in the absence of disease progression
  Arms: Arm A
Drug: Placebo — 20mg od (continuous dosing) until evidence of disease progression has been confirmed
  Arms: Arm A
Drug: cisplatin — cisplatin 25 mg/m2 on days 1 and 8 of a 21-day cycle for 24 weeks in the absence of disease progression
  Arms: B
Drug: cediranib — cediranib 20mg oral daily (continuous dosing)until evidence of disease progression has been confirmed
  Other Names: AZD2171
  Arms: B
Drug: gemcitabine — gemcitabine 1000 mg/m2 on days 1 and 8 of a 21-day cycle for 24 weeks in the absence of disease progression
  Arms: B

SUMMARY:
As a result of our previous NCRN study (ABC-02) cisplatin and gemcitabine (CisGem) is likely to become the international standard of care for patients with advanced biliary tract cancer (submitted: ASCO 2009).

This study, ABC-03, will determine whether the addition of cediranib(an oral Vascular Endothelial Growth Factor Receptor inhibitor) to CisGem will improve the time to disease progression in this patient group.

DETAILED DESCRIPTION:
Although there is currently no standard chemotherapy for patients with advanced biliary tract cancers (ABC) the UK ABC-02 study (the largest study by far in this patient group, n=410) is likely to define CisGem as the global standard of care for this disease based on a significantly improved progression-free survival and overall survival compared to gemcitabine alone.

Vascular endothelial growth factor (VEGF) is a pivotal stimulus of physiologic and pathologic angiogenesis, including the sustained neo-vascularisation required to support solid tumour growth. Human biliary tract carcinoma cells have higher expression of VEGF both in cell lines and tissues (detected in 75.6% of 33 resected clinical specimens) and this is associated with significantly higher levels of microvessel density and the presence of intrahepatic metastases.

Cediranib is a highly potent inhibitor of VEGF receptor 2 tyrosine kinase and VEGF-induced signalling in endothelial cells. It has been safely combined with a CisGem regimen in lung cancer patients.

Aims This trial aims to evaluate the effect on progression-free survival of cediranib in combination with CisGem chemotherapy compared to CisGem and placebo.

Summary of study Consenting patients with ABC (inoperable, locally advanced, recurrent or metastatic) will receive CisGem chemotherapy and either cediranib (experimental arm) or placebo (standard arm) orally. Treatment will continue until disease progression (chemotherapy will stop at 24 weeks) with tumour reassessment by CT/MRI scans at 12-weekly intervals. All patients will be followed up for survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* A histopathological/cytological diagnosis of non-resectable or recurrent/metastatic biliary tract carcinoma (intra- or extra-hepatic), gallbladder or ampullary carcinoma
* Measurable disease on CT or MR scanning. Radiological assessments must be done within 4 weeks of randomisation
* ECOG performance status 0 or 1
* Age ≥ 18 and estimated life expectancy > 3 months
* Adequate haematological function: Haemoglobin ≥ 10g/dl*; WBC ≥ 3.0 x 109/L; Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelet count ≥ x 109/L, *prior transfusions for patients with low haemoglobin are allowed
* Adequate liver function : Total bilirubin ≤1.5 x upper limit of normal (ULN); ALT and/or AST ≤ 2.5 x ULN (If liver metastases are present, ALT or AST < 5 x ULN)
* Alkaline phosphatase ≤ 5 x ULN
* Adequate renal function with serum urea and serum creatinine < 1.5 times ULN and a calculated GFR ≥ 45 mL/min. If the calculated GFR is below 45 mL/min, isotope EDTA confirmation of adequate renal function is required
* Adequate biliary drainage, with no evidence of active uncontrolled infection (patients on long-term antibiotics are eligible provided signs of active infection have resolved)
* Women of child-bearing potential should have a negative pregnancy test prior to study entry AND be using an adequate contraception method, which must be continued for 3 months after completion of chemotherapy

Exclusion Criteria:

* Significant haemorrhage (>30 mL bleeding/episode in previous 3 months) or haemoptysis (>5 mL fresh blood in previous 4 weeks)
* Patients with history of poorly controlled hypertension with resting blood pressure >150/100 mmHg in the presence or absence of a stable regimen of anti-hypertensive therapy, or patients who are requiring maximal doses of calcium channel blockers to stabilise blood pressure
* Incomplete recovery (grade CTC >1) from previous anti-cancer therapy (except haematological toxicity - see eligibility for adequate haematological function, or alopecia) or unresolved biliary tree obstruction
* Prior therapy with chemoradiotherapy (either adjuvant or in the locally advanced setting)
* Any evidence of severe or uncontrolled systemic diseases which, in the view of the investigator, makes it undesirable for the patient to participate in the trial (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
* Untreated unstable brain or meningeal metastases. Patients with radiological evidence of stable brain metastases are eligible providing that they are asymptomatic and either do not require corticosteroids or have been treated with corticosteroids, with clinical and radiological evidence of stabilisation at least 10 days after discontinuation of steroids
* Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart unless urinary protein <1.5 g in a 24-hour period
* History of significant gastrointestinal impairment, as judged by the Investigator, that would significantly affect the absorption of cediranib
* Mean QTc with Bazetts correction >470 msec in screening ECG or history of familial long QT syndrome
* Recent (<14 days) major thoracic or abdominal surgery prior to entry into the study, or a surgical incision that is not fully healed
* Pregnant or breast-feeding women or women of childbearing potential with a positive pregnancy test prior to receiving study medication
* Known hypersensitivity to cediranib or any of its excipients
* Known risk of the patient transmitting HIV, hepatitis B or C via infected blood
* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site(s)
* Previous enrolment or randomisation of treatment in the present study
* Treatment with an investigational (non-registered) drug within 30 days prior to the first dose of cediranib
* Other concomitant anti-cancer therapy (except steroids)
* Incomplete recovery from previous surgery or unresolved biliary tract obstruction
* Patients undergoing current treatment with curative intent
* History of prior malignancy that will interfere with the response evaluation (exceptions include in-situ carcinoma of the cervix treated by cone-biopsy/resection, non-metastatic basal and/or squamous cell carcinomas of the skin, any early stage (stage I) malignancy adequately resected for cure greater than 5 years previously)
* Any evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial
* Any psychiatric or other disorder (eg brain metastases) likely to impact on informed consent
* NB. Whilst not excluded, patients with significant impaired hearing must be made aware of potential ototoxicity and may choose not to be included. If included, it is recommended that audiograms be carried out at baseline and prior to cycle 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival | six months

SECONDARY OUTCOMES:
• Response Rate (RECIST) • Toxicity • Survival (as part of the follow-on phase III study) • Biomarker evaluation (inc. circulating VEGF, sVEGFR-2, bFGF, LDH and CA 19-9) • Quality of Life | 3 years minimum

CONTACTS AND LOCATIONS:
Overall Officials: Juan Valle, MD, Principal Investigator — The Christie NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Valle JW, Wasan H, Lopes A, Backen AC, Palmer DH, Morris K, Duggan M, Cunningham D, Anthoney DA, Corrie P, Madhusudan S, Maraveyas A, Ross PJ, Waters JS, Steward WP, Rees C, Beare S, Dive C, Bridgewater JA. Cediranib or placebo in combination with cisplatin and gemcitabine chemotherapy for patients with advanced biliary tract cancer (ABC-03): a randomised phase 2 trial. Lancet Oncol. 2015 Aug;16(8):967-78. doi: 10.1016/S1470-2045(15)00139-4. Epub 2015 Jul 12. PMID 26179201